CLINICAL TRIAL: NCT01904617
Title: A Randomized Controlled Trial on the Effects of Rate and/or Presence of Dextrose on the Labor Course of Nulliparas
Brief Title: Effects of Rate and/or Presence of Dextrose on the Labor Course of Nulliparas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 025-11
Record Dates: First submitted 2013-04-19; First posted 2013-07-22 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Length of Labor; Second Stage of Labor; Intravenous Hydration of Labor
Keywords: Length of labor; second stage of labor; intravenous hydration of labor; intravenous glucose
MeSH Terms: interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- D5NS at 125 mL/hr (Experimental): 5% dextrose in normal saline at 125 mL/hr
  Interventions: Other: Dextrose; Other: Normal Saline
- D2.5NS at 250mL/hr (Experimental): 2.5% dextrose in normal saline at 250 mL/hr
  Interventions: Other: Dextrose; Other: Normal Saline
- NS at 250mL/hr (Experimental): Normal saline at 250mL/hr
  Interventions: Other: Normal Saline

INTERVENTIONS:
Other: Dextrose
  Arms: D2.5NS at 250mL/hr; D5NS at 125 mL/hr
Other: Normal Saline
  Other Names: Intravenous fluids, normal saline

SUMMARY:
This randomized controlled trial aims to compare three groups of intravenous fluids and their impact on labor: 1) 125 mL/hr of 5% dextrose in normal saline 2) 250 mL/hr of normal saline 3) 250 mL/hr of 5% dextrose in normal saline

DETAILED DESCRIPTION:
Currently, patients who arrive to labor and delivery automatically receive IV fluid hydration as part of a standard order set. The current default IV fluid order is 125mL/hr of 5% dextrose, either in normal saline or lactated ringers.

Any patient delivering for the first time presenting to labor and delivery in active labor will be screened. If they meet inclusion requirements they will be offered enrollment.

Subjects will be blindly randomized to receive one of three different types of IV fluids:

1. 5% dextrose Normal saline (Normal saline plus 5g/dl of glucose) at 125 mL/hr (the current LBMMC default inpatient IV order set)
2. Normal saline (a solution containing sodium and chloride) at 250 mL/hr
3. 2.5% dextrose Normal saline at 125 mL/hr

   * Management of labor will be at the discretion of the attending physician(s).
   * Maternal outcomes to be measured include: 1) total amount of IV fluids administered, 2) length of labor, 3) epidural use, 4) oxytocin use, 5) mode of delivery, 6) development of maternal infections or other morbidity such as postpartum hemorrhage.
   * Neonatal outcomes to be measured include: 1) birth weight, 2) Apgar scores, 3) hospital course (nursery placement and length of stay), 4) need for treatment of jaundice.

ELIGIBILITY:
Inclusion Criteria:

* • Primiparous

  * Singleton gestation
  * Vertex presentation
  * Spontaneous active labor with or without pitocin augmentation
  * Gestational age > 36 weeks
  * Cervical dilation 3 to 5 cm with or without ruptured membranes

Exclusion Criteria:

* • Multiparous

  * Pregestational or gestational diabetes mellitus
  * Preeclampsia at admission
  * Previous cesarean section
  * Non-vertex presentation
  * Multiple gestation
  * Chorioamnionitis at admission
  * Intrauterine growth restriction (< 10th percentile)
  * Patients admitted for induction
  * BMI > 50

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Length of labor | Time from fluid initiation to delivery

SECONDARY OUTCOMES:
Time of second stage of labor | Time from initiation of pushing to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Vineet Shrivastava, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States